CLINICAL TRIAL: NCT06773195
Title: A Phase 1/2 Study of Combined JAK/ERK Inhibition in Patients With Myelofibrosis
Brief Title: A Study of Ruxolitinib in Combination With Ulixertinib in People With Myelofibrosis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: BioMed Valley Discoveries, Inc (Industry); Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-157
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Myelofibrosis
Keywords: post-ET myelofibrosis; post-PV myelofibrosis,; post-pre-fibrotic myelofibrosis; JAK/MEK inhibition; Ruxolitinib; Ulixertinib
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ulixertinib; ruxolitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JAK/MEK inhibition with Ruxolitinib and Ulixertinib (Experimental): Phase 1: There are 3 planned dose levels of ulixertinib (450 mg BID, 300 mg BID, or 150 mg BID) in combination with ruxolitinib for 28 day cycles. A 3+3 dose escalation design will be used to determine the RP2D of ulixertinib with ruxolitinib. Phase 2: Participants will be treated with ulixertinib at the RP2D determined from the phase 1 part of the study in combination with ruxolitinib for 28 day cycles.
  Interventions: Drug: Ulixertinib; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ulixertinib — There are 3 planned dose levels of ulixertinib(450 mg BID, 300 mg BID, or 150 mg BID)
Drug: Ruxolitinib — Ruxolitinib for 28 day cycles.

SUMMARY:
The researchers are doing this study to find out whether the combination of ruxolitinib and ulixertinib is a safe and effective treatment for people with myelofibrosis. The researchers will test different doses of ulixertinib to find the highest dose that causes few or mild side effects in participants when given in combination with ruxolitinib.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of primary myelofibrosis, post-ET myelofibrosis, post-PV myelofibrosis, or post-pre-fibrotic myelofibrosis by WHO 2016 criteria.
* Age ≥18 years.
* Receiving ruxolitinib monotherapy for at least 3 months with stable dose (10 mg BID to 20mg BID) for at least 4 weeks before first dose of study drug. Note: stable ruxolitinib dosing should be achieved according to strict adherence to dose modification/reduction guidelines detailed in the ruxolitinib package insert, for patients with renal impairment, and/or hepatic impairment.
* Must have DIPSS+ intermediate 2 or greater risk disease, or MIPSS70+ intermediate or greater risk disease
* Persistent disease despite ruxolitinib monotherapy, as demonstrated by:

  o Grade 2 or 3 reticulin/collagen fibrosis on bone marrow AND
  * Splenomegaly (palpable at least 5cm below subcostal margin/or spleen volume > 450cm^3) OR
  * Active symptoms (MPN-SAF TSS score >10 with at least one MPNSAF TSS score >5 or two scores >3) OR
* ECOG performance status ≤2
* Participants must have adequate organ and marrow function as defined below unless the elevated laboratory values are attributable to Gilbert's Syndrome with Sponsor review and approval:

  * Absolute neutrophil count ≥ 0.5 K/mcL
  * Platelets ≥ 50 K/mcL
  * Direct bilirubin ≤ 1.5 times institutional upper limit of normal (ULN)
  * Total bilirubin ≤ 1.5 times institutional upper limit of normal (ULN
  * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN
  * Creatinine clearance ≥ 50 mL/min as calculated by institutional standard
  * Bone marrow and peripheral blood blast count <10%
* Agreeable to the use of adequate contraception to avoid pregnancy (Appendix D). Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth contro) prior to study entry, for the duration of study participation, and 4 months after completion of drug administration (Appendix D). At least two highly effective methods of contraception, one of which must be a barrier method, are required for males and females of childbearing age during dosing and for 4 months after completing treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of drug administration

Exclusion Criteria:

* Use of experimental drug therapy for MF or any other standard drug with the exception of hydroxyurea or ruxolitinib within 2 weeks of starting combination therapy and/or lack of recovery from all toxicities from previous therapy (except ruxolitinib) to Grade 1 or better. Hydroxyurea may be utilized to control leukocytosis for up to 4 weeks during study
* Participants with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Unwilling to receive red blood cell transfusion to treat low hemoglobin.
* Participants who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ruxolitinib and ulixertinib.
* Participants requiring any medications or substances that are strong inhibitors or inducers of 3A4, strong inhibitors of CYP1A2 and CYP2D6, and inhibitors of Pglycoprotein (P-gp). Strong inhibitors or inducers of 3A4, strong inhibitors of CYP1A2 and CYP2D6, and inhibitors of P-gp must be stopped within 14 days (or 5 half-lives) of study commencement. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.
* Participants who are pregnant or breastfeeding.
* Pregnant women are excluded from this study because ruxolitinib and ulixertinib are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ruxolitinib and ulixertinib, breastfeeding should be discontinued if the mother is treated with ruxolitinib and ulixertinib.
* Active bacterial, fungal, or viral infection requiring treatment.
* Participants with chronic Human immunodeficiency virus (HIV) or hepatitis B or C viral infection.

  * HIV-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial. Note: testing does not have to be performed during screening unless participant has known or suspected history of HIV.
  * For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Presence of active interstitial lung disease or pneumonitis.
* History of cardiovascular risk factors:

  * Clinically significant, uncontrolled arrythmias and/or conduction abnormalities. Participants with controlled atrial fibrillation >30 days prior to study initiation are eligible.
  * QTc > 480 msec.
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to study entry;
  * Class II congestive heart failure or greater or ejection fraction ≤50% on baseline echocardiogram.
  * History of uncontrolled hypertension.
* A history or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR).
* Psychiatric illness/social situations, active drug, alcohol or substance use that would interfere with study compliance.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending study visits; pose a significant risk to the participant; or interfere with interpreting study data.
* Participants eligible for allogeneic stem cell transplantation in the opinion of the treating physician at the time of enrollment.
* Inability to comprehend or unwilling to sign the informed consent form.
* Transformation to accelerated or blast phase disease, including myeloid sarcoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity evaluable participants | up to 28 days
  If none of the initial 3 patients in a cohort experience a dose limiting toxicity (DLT), then the next dose level will be studied in another cohort of 3 patients. If 1 of the initial 3 patients at a given dose level experience a DLT, up to 3 additional patients will be treated at that same dose level. Escalation will continue if not more than 1 of the 6 patients experience a DLT.
Response to therapy | at week 25
  as defined by International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT working criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Raajit Rampal, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - Massachusetts General Hospital (Data Collection Only), Boston, Massachusetts
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm